CLINICAL TRIAL: NCT06892808
Title: Effectiveness of Non-Surgical Periodontal Therapy on Atrial Fibrillation Recurrence After Radiofrequency Ablation in Patients with Atrial Fibrillation and High-Inflammatory Burden Periodontitis
Brief Title: Impact of Periodontal Therapy on AF Recurrence Post-Ablation in High-Inflammatory Burden Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xu Liu (Other)
Collaborators: The First People's Hospital of Hefei City (Unknown); The Second People's Hospital of Anhui Province (Other)
Responsible Party: Sponsor-Investigator, Xu Liu, Professor, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIPDAF
Record Dates: First submitted 2025-03-02; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation; Periodontitis
Keywords: Atrial Fibrillation; Periodontitis
MeSH Terms: conditions — Atrial Fibrillation; Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Non-Surgical Periodontal Therapy Protocol Under local anesthesia, full-mouth debridement (supragingival and subgingival scaling and root planing, FM-SRP) was performed by an experienced periodontist, initiated within 48 hours post-atrial fibrillation ablation and completed in two sessions within 48 hours. Polishing was performed using a rubber cup with prophylaxis paste. The procedure utilized Gracey curettes and piezoelectric ultrasonic tips combined with a force-controlled system.
  Postoperative Care Immediate Care:Local Adjunctive Therapy: 2% minocycline gel was injected into deep periodontal pockets (PD ≥5mm). Antimicrobial Rinse: 0.12% chlorhexidine solution (15 mL, 30-second rinse twice daily) for 14 days.
  Follow-Up Intervention At the 6-month follow-up, additional oral debridement was performed in the intervention group if indicated by the presence of bleeding points and/or increased probing pocket depth (PPD).
  Interventions: Procedure: Non-Surgical Periodontal Therapy; Procedure: Background Periodontal Care
- Control group (Active Comparator): All study participants received oral hygiene instruction using the modified Bass technique. At baseline, supragingival deposits (dental plaque and calculus) were removed with an ultrasonic scaler or rubber cup with prophylaxis paste. To maintain blinding, simulated subgingival instrumentation sounds were played during the procedure for control group participants.
  Interventions: Procedure: Background Periodontal Care

INTERVENTIONS:
Procedure: Non-Surgical Periodontal Therapy — Under local anesthesia, full-mouth debridement (supragingival and subgingival scaling and root planing, FM-SRP) was performed by an experienced periodontist, initiated within 48 hours post-atrial fibrillation ablation and completed in two sessions within 48 hours. Polishing was performed using a rubber cup with prophylaxis paste. The procedure utilized Gracey curettes and piezoelectric ultrasonic tips combined with a force-controlled system.
  Postoperative Care Immediate Care: Local Adjunctive Therapy: 2% minocycline gel was injected into deep periodontal pockets (PD ≥5mm). Antimicrobial Rinse: 0.12% chlorhexidine solution (15 mL, 30-second rinse twice daily) for 14 days.
  Follow-Up Intervention At the 6-month follow-up, additional oral debridement was performed in the intervention group if indicated by the presence of bleeding points and/or increased probing pocket depth (PPD).
  Arms: Treatment group
Procedure: Background Periodontal Care — All study participants received oral hygiene instruction using the modified Bass technique. At baseline, supragingival deposits (dental plaque and calculus) were removed with an ultrasonic scaler or rubber cup with prophylaxis paste. To maintain blinding, simulated subgingival instrumentation sounds were played during the procedure for control group participants.

SUMMARY:
Comparison of Non-Surgical Periodontal Therapy versus Background Periodontal Care in Reducing Atrial Fibrillation Recurrence in Patients with AF and Periodontitis: A Randomized Trial with Two Arms (Background Therapy Group vs. Conventional Non-Surgical Therapy Group).

ELIGIBILITY:
Inclusion Criteria:

- Age ≥18 years. Diagnosed with atrial fibrillation (AF) and undergoing first-time catheter ablation.

Diagnosed with periodontitis (2017 World Workshop classification) and periodontal inflamed surface area (PISA) >500 mm².

Willing and able to provide written informed consent.

Exclusion Criteria:

- Requiring periodontal surgical intervention, e.g., flap surgery, bone grafting. Non-surgical periodontal therapy (e.g., scaling and root planing) within the past 6 months.

Active systemic infection, e.g., sepsis, tuberculosis. Current immunosuppressive therapy, e.g., post-transplant medications, long-term corticosteroids.

Chronic hepatitis B or HIV infection. Chronic systemic antibiotic use (>4 weeks). Pregnancy or lactation. Anticipated survival <12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation (AF) episodes lasting ≥30 seconds occurring | From 3 months post-ablation (end of blanking period) to the 12-month follow-up.
  Atrial fibrillation (AF) episodes lasting ≥30 seconds occurring from 3 months post-ablation (end of blanking period) to the 12-month follow-up.

SECONDARY OUTCOMES:
Composite atrial arrhythmia recurrence | During the period from 3 months post-ablation to 12-month follow-up.
  AF, atrial flutter (AFL), or atrial tachycardia (AT) episodes lasting ≥30 seconds during the period from 3 months post-ablation to 12-month follow-up.
Antiarrhythmic drug usage | At 12 months.
  Antiarrhythmic drug usage at 12 months.
Change in Periodontal Inflamed Surface Area (PISA) | At 12 months
  Change in Periodontal Inflamed Surface Area (PISA) at 12 months
Probing depth (PD) reduction ≥2 mm in ≥50% of sites. | At 12 months.
  Probing depth (PD) reduction ≥2 mm in ≥50% of sites.
Bleeding on probing (BOP) rate reduction ≥30%. | At 12 months.
  Bleeding on probing (BOP) rate reduction ≥30%.
Clinical attachment level (CAL) stability (change ≤1 mm). | At 12 months.
  Clinical attachment level (CAL) stability (change ≤1 mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Xuhui, China

IPD SHARING:
Plan to Share IPD: No